CLINICAL TRIAL: NCT01809366
Title: Effect of Seminal Plasma Insemination on Pregnancy Rates After IVF-ET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Senior, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 65/10
Record Dates: First submitted 2013-03-10; First posted 2013-03-12 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-01

CONDITIONS: Effect on Implantation and Pregnancy Rates
Keywords: seminal plasma/uterine receptivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- seminal plasma insemination (Experimental): seminal plasma insemination
  Interventions: Procedure: seminal plasma insemination
- culture medium insemination (Placebo Comparator): culture medium insemination
  Interventions: Procedure: seminal plasma insemination

INTERVENTIONS:
Procedure: seminal plasma insemination

SUMMARY:
Seminal plasma insemination into the vaginal vault of patients undergoing IVF-ET increases uterine receptivity.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing oocyte pick up for IVF treatment

Exclusion Criteria:

* endometriosis
* low responders
* uterine malformations

Ages: 20 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2012-01; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
implantation rate | 4 weeks after ET

SECONDARY OUTCOMES:
clinical pregnancy rate | 4 weeks after ET
ongoing pregnancy rate | 6 weeks after ET

CONTACTS AND LOCATIONS:
Locations (1):
- Infertility and IVF Unit, Assaf harofeh Medical Center, Zrifin, Israel